CLINICAL TRIAL: NCT00683878
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Combination With Thiazolidinedione Therapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Thiazolidinedione Therapy Alone
Brief Title: Add-on to Thiazolidinedione (TZD) Failures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Astra Zeneca, Bristol-Myers Squibb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB102-030
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; 2,4-thiazolidinedione; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Thiazolidinedione (Pioglitazone)
- Arm 2 (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Thiazolidinedione (Pioglitazone)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo matching Dapagliflozin; Drug: Thiazolidinedione (Pioglitazone)

INTERVENTIONS:
Drug: Dapagliflozin — Tablets, Oral, 5.0 mg, once daily, up to 48 weeks
  Other Names: BMS-512148
  Arms: Arm 1
Drug: Dapagliflozin — Tablets, Oral, 10.0 mg, once daily, up to 48 weeks
  Other Names: BMS-512148
  Arms: Arm 2
Drug: Placebo matching Dapagliflozin — Tablets, Oral, 0 mg, once daily, up to 48 weeks
  Arms: Arm 3
Drug: Thiazolidinedione (Pioglitazone) — Tablets, ≥ 30 mg, Once daily, up to 48 weeks

SUMMARY:
The purpose of this clinical research study is to learn if BMS-512148 (Dapagliflozin) can help reduce the blood sugar levels in subjects with Type 2 Diabetes who are not well controlled on TZD alone. The safety of this treatment will also be studied

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥ 18 years old, with type 2 diabetes and with inadequate glycemic control
* All subjects must have central laboratory pre-randomization A1C ≥ 7.0 and ≤ 10.5%
* C-peptide ≥ 1.0 ng/mL (0.34 nmol/L)
* Body Mass Index ≤ 45.0 kg/m²

Exclusion Criteria:

* AST and /or ALT > 2.5 times the upper limit of normal
* Serum total bilirubin > 2 mg/dL (34.2 µmol/L)
* Creatinine kinase > 3.0 times the upper limit of normal
* Symptoms of severely uncontrolled diabetes
* Serum creatinine ≥ 2.0 mg/dL
* Calculated Cr-Clearance < 50 ml/min (calculated by Cockroft-Gault formula)
* Currently unstable or serious cardiovascular, renal, hepatic, hematological, oncological, endocrine, psychiatric, or rheumatic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 972 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (86):
- United States (57):
  - Pinnacle Research Group, Llc, Anniston, Alabama
  - Iicr, Ozark, Alabama
  - 43rd Medical Associates, P.C., Phoenix, Arizona
  - Clinical Research Advantage Inc / Desert Clinical Res, Llc, Tempe, Arizona
  - Clinical Research Advantage, Inc, Tempe, Arizona
  - Little Rock Family Practice Clinic, Little Rock, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - Clinical Innovations, Inc., Costa Mesa, California
  - Marin Endocrine Care And Research, Inc., Greenbrae, California
  - Torrance Clinical Research, Lomita, California
  - Randall Shue, D.O., Los Angeles, California
  - Diabetes Medical Center Of California, Northridge, California
  - Desert Medical Advances, Palm Desert, California
  - Avastra Clinical Trials, Redlands, California
  - Sierra Clinical Research, Roseville, California
  - Ritchken & First M.D.'S, San Diego, California
  - Advantage Clinical Research, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Diabetes Research Center, Tustin, California
  - Aurora Family Medicine Center, P.C., Aurora, Colorado
  - Denver Internal Medicine, Denver, Colorado
  - Central Florida Clinical Trials, Altamonte Springs, Florida
  - Health First Clinical Research Group, Inc., Chipley, Florida
  - Clinical Therapeutics Corporation, Coral Gables, Florida
  - Westside Center For Clinical Research, Jacksonville, Florida
  - Panhandle Family Care Associates, Marianna, Florida
  - Baptist Diabetes Associates, Pa, Miami, Florida
  - Suncoast Clinical Res Inc., New Port Richey, Florida
  - Stone Mountain Clinical Research, Stone Mountain, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Northwest Indiana Center For Clinical Research, Valparaiso, Indiana
  - Professional Research Network Of Kansas, Wichita, Kansas
  - St. Mary'S Center For Diabetes And Endocrinology, Grand Rapids, Michigan
  - Endocrine Research Associates, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Danny W. Jackson P.A., Rolling Fork, Mississippi
  - Association Of International Professionals, Las Vegas, Nevada
  - Physicians Research Center, Toms River, New Jersey
  - Finger Lakes Clinical Research, Rochester, New York
  - Metrolina Internal Medicine, Charlotte, North Carolina
  - The Center For Nutrition & Preventive Medicine, Pllc, Charlotte, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Providence Health Partners - Center For Clinical Research, Dayton, Ohio
  - Physician Research, Inc., Zanesville, Ohio
  - Family Medical Associates, Levittown, Pennsylvania
  - Banksville Medical, Pc, Pittsburgh, Pennsylvania
  - Brookside Family Practice & Pediatrics, Pottstown, Pennsylvania
  - Columbia Clinical Research, Inc., Columbia, South Carolina
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Dallas Diabetes & Endocrine Center, Dallas, Texas
  - Village Family Practice, Houston, Texas
  - Office Of Dr. Michelle Zaniewski Singh, Houston, Texas
  - Diabetes & Glandular Disease Research Assoc,, Inc., San Antonio, Texas
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - William L. Gray, Md, Spokane, Washington
- Argentina (4):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Ciudad Auton, Buenos Aires
  - Local Institution, Zárate, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
- Canada (7):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Sarnia, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Mirabel, Quebec
- India (3):
  - Local Institution, Hariyāna
  - Local Institution, Mumbai
  - Local Institution, Vellore
- Mexico (7):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Monterrey, Nl, Nuevo León
  - Local Institution, Veracruz, Veracruz
  - Local Institution, Mérida, Yucatán
- Local Institution, Lima, Lima Province, Peru
- Philippines (3):
  - Local Institution, Cebu City
  - Local Institution, Manila
  - Local Institution, Pasig
- Local Institution, Ponce, Puerto Rico
- Taiwan (3):
  - Local Institution, Changhua
  - Local Institution, Taichung
  - Local Institution, Taipei

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Shah M, Stolbov L, Yakovleva T, Tang W, Sokolov V, Penland RC, Boulton D, Parkinson J. A model-based approach to investigating the relationship between glucose-insulin dynamics and dapagliflozin treatment effect in patients with type 2 diabetes. Diabetes Obes Metab. 2021 Apr;23(4):991-1000. doi: 10.1111/dom.14305. Epub 2021 Jan 25. PMID 33368935
- [Derived] Kohan DE, Fioretto P, Johnsson K, Parikh S, Ptaszynska A, Ying L. The effect of dapagliflozin on renal function in patients with type 2 diabetes. J Nephrol. 2016 Jun;29(3):391-400. doi: 10.1007/s40620-016-0261-1. Epub 2016 Feb 19. PMID 26894924
- [Derived] Rosenstock J, Vico M, Wei L, Salsali A, List JF. Effects of dapagliflozin, an SGLT2 inhibitor, on HbA(1c), body weight, and hypoglycemia risk in patients with type 2 diabetes inadequately controlled on pioglitazone monotherapy. Diabetes Care. 2012 Jul;35(7):1473-8. doi: 10.2337/dc11-1693. Epub 2012 Mar 23. PMID 22446170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 972 participants enrolled, 558 completed a qualification period. Before entering lead-in period, 344 participants entered dose optimization period and 263 completed. A total of 480 participants entered the lead-in period, 420 randomized and received treatment, 367 completed double-blind treatment period.
Groups:
- PLACEBO + Pioglitazone: Placebo tablets, oral, once daily, up to 48 weeks plus pioglitazone tablets, ≥ 30 mg, once daily up to 48 weeks
- Dapagliflozin 5MG + Pioglitazone; Dapagliflozin 10MG + Pioglitazone: Dapagliflozin tablets, oral, once daily, up to 48 weeks plus pioglitazone tablets, ≥ 30 mg, once daily up to 48 weeks
Period: Overall Study
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Started | 139 | 141 | 140
Completed | 116 | 125 | 126
Not Completed | 23 | 16 | 14
Not completed — Lack of Efficacy | 3 | 0 | 1
Not completed — Adverse Event | 4 | 3 | 3
Not completed — Withdrawal by Subject | 9 | 8 | 6
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 2 | 4
Not completed — Non-compliance, not met criteria etc. | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone | Total
Number analyzed (Participants) | 139 | 141 | 140 | 420
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (11.38) | 53.2 (10.90) | 53.8 (10.35) | 53.5 (10.86)
Age, Customized [Number; unit: Participants]
  Yonger than 65 years | 115 | 120 | 118 | 353
  65 to younger than 75 years | 21 | 16 | 20 | 57
  75 years and older | 3 | 5 | 2 | 10
Gender [Count of Participants; unit: Participants]
  Female | 68 | 63 | 81 | 212
  Male | 71 | 78 | 59 | 208
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 24 | 26 | 21 | 71
  Black/African American | 6 | 9 | 7 | 22
  White | 102 | 102 | 101 | 305
  Other | 7 | 4 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hemoglobin A1C (HbA1c) at Week 24 (Last Observation Carried Forward [LOCF])
Description: HbA1c was measured as percent of hemoglobin by a central laboratory. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. HbA1c measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing HbA1c values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: % of hemoglobin
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 138 | 140 | 140
% of hemoglobin | -0.42 (0.0834) | -0.82 (0.0828) | -0.97 (0.0828)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; p = 0.0007, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.63 to -0.17], Standard Error of Mean 0.1175
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Primary endpoints were tested at alpha=0.027 applying Dunnett's adjustment; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.78 to -0.31], Standard Error of Mean 0.1175

2. Secondary Outcome: Adjusted Mean Change From Baseline in 120-minute Post-challenge Plasma Glucose (PPG) (mg/dL) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. In post oral glucose tolerance test (OGTT), glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. PPG measurements were obtained on Day 1 and week 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 112 | 116 | 115
mg/dL | -14.1 (6.421) | -65.1 (6.325) | -67.5 (6.359)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -51.0, 95% CI 2-sided [-68.7 to -33.2], Standard Error of Mean 9.007
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -53.3, 95% CI 2-sided [-71.1 to -35.6], Standard Error of Mean 9.039

3. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing body weight values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: kg
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 139 | 140 | 140
kg | 1.64 (0.2760) | 0.09 (0.2752) | -0.14 (0.2753)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-2.32 to -0.79], Standard Error of Mean 0.3896
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.78, 95% CI 2-sided [-2.55 to -1.02], Standard Error of Mean 0.3896

4. Secondary Outcome: Adjusted Mean Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Fasting plasma glucose was measured as milligrams per deciliter(mg/dL) by a central laboratory. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. FPG measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 in the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing FPG values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 139 | 140 | 140
mg/dL | -5.5 (2.893) | -24.9 (2.884) | -29.6 (2.880)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -19.5, 95% CI 2-sided [-27.5 to -11.4], Standard Error of Mean 4.088
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -24.1, 95% CI 2-sided [-32.2 to -16.1], Standard Error of Mean 4.082

5. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response (Hemoglobin A1c [HbA1C]) <7.0% at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Percent adjusted for baseline HbA1c. Therapeutic glycemic response is defined as HbA1c <7.0%. Data after rescue medication was excluded from this analysis. HbA1c was measured as a percent of hemoglobin. Mean and standard error for percentage of participants were estimated by modified logistic regression model.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: Percentage of participants
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 138 | 140 | 140
Percentage of participants | 22.4 (3.276) | 32.5 (3.669) | 38.8 (3.835)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; p = 0.0496, Modified logistic regression — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [0.0 to 20.1], Standard Error of Mean 5.119
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p = 0.0018, Modified logistic regression — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = 16.4, 95% CI 2-sided [6.1 to 26.7], Standard Error of Mean 5.253

6. Secondary Outcome: Adjusted Mean Change From Baseline in Waist Circumference (cm) at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in waist circumference at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Waist circumference measurements were obtained during the qualification and lead-in periods and on Day 1 and Week 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing waist circumference values at baseline and Week 24 (LOCF)
Measure: Mean (Standard Error); unit: cm
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 126 | 132 | 133
cm | 1.38 (0.4301) | 0.52 (0.4198) | -0.17 (0.4182)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; p = 0.1566, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -0.85, 95% CI 2-sided [-2.03 to 0.33], Standard Error of Mean 0.6006
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p = 0.0101, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-2.73 to -0.37], Standard Error of Mean 0.5995

7. Secondary Outcome: Adjusted Mean Change From Baseline in Total Body Weight (kg) Among Subjects With Baseline Body Mass Index (BMI) ≥ 27 kg/m^2 at Week 24 (Last Observation Carried Forward [LOCF])
Description: Secondary endpoints were tested using sequential testing procedure and are presented in hierarchical order. Adjusted mean change from baseline in total body weight among subjects with baseline body mass index (BMI) ≥ 27 kg/m^2 at Week 24 (or the last postbaseline measurement prior to Week 24 if no Week 24 assessment was available was determined. Data after rescue medication was excluded from this analysis. Baseline was defined as the last assessment prior to the start date and time of the first dose of the double-blind study medication. In cases where time of the first dose or time of the assessment was not available, baseline was defined as the last assessment on or prior to the date of the first dose of the double-blind study medication. Body weight measurements were obtained during the qualification and lead-in periods and on Day 1 and Weeks 1, 2, 4, 8, 12, 16, 20, and 24 of the double-blind period.
Time Frame: From Baseline to Week 24
Population: All randomized participants who received study medication and had nonmissing body weight values at baseline and Week 24 (LOCF) among subjects with baseline body mass index (BMI) ≥ 27 kg/m^2
Measure: Mean (Standard Error); unit: kg
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Number analyzed (Participants) | 113 | 101 | 113
kg | 1.83 (0.3313) | 0.26 (0.3523) | -0.07 (0.3332)
Statistical Analysis 1: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 5MG + Pioglitazone; Test type: Superiority or Other; ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05. The comparison was stopped due to the preceding test (PLACEBO + Pio vs Dapa 5MG + Pio) not statistically significant P value = 0.1566; Mean Difference (Final Values) = -1.58, 95% CI 2-sided [-2.53 to -0.62], Standard Error of Mean 0.4838
Statistical Analysis 2: Comparison: PLACEBO + Pioglitazone vs Dapagliflozin 10MG + Pioglitazone; Test type: Superiority or Other; p < 0.0001, ANCOVA — Secondary endpoints were tested following a sequential testing procedure at alpha=0.05; Mean Difference (Final Values) = -1.90, 95% CI 2-sided [-2.83 to -0.98], Standard Error of Mean 0.4688

ADVERSE EVENTS:
Time Frame: Onset on or after the first date of double-blind treatment and on or prior to the last day of double-blind treatment 24 weeks plus 4 days for non-serious adverse event; plus 30 days for serious adverse event.
Arm/Group | PLACEBO + Pioglitazone | Dapagliflozin 5MG + Pioglitazone | Dapagliflozin 10MG + Pioglitazone
Serious Adverse Events (participants affected / at risk) | 1/139 | 4/141 | 2/140
Other Adverse Events (participants affected / at risk) | 37/139 | 34/141 | 45/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO + Pioglitazone (N=139) | Dapagliflozin 5MG + Pioglitazone (N=141) | Dapagliflozin 10MG + Pioglitazone (N=140)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO + Pioglitazone (N=139) | Dapagliflozin 5MG + Pioglitazone (N=141) | Dapagliflozin 10MG + Pioglitazone (N=140)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 6 (7) | 8 (8) | 13 (14)
NASOPHARYNGITIS (Infections and infestations) | 5 (7) | 7 (7) | 11 (11)
DIARRHOEA (Gastrointestinal disorders) | 6 (7) | 4 (4) | 9 (9)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5) | 7 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 9 (11) | 7 (8)
HEADACHE (Nervous system disorders) | 9 (9) | 3 (4) | 4 (4)
OEDEMA PERIPHERAL (General disorders) | 7 (7) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No